CLINICAL TRIAL: NCT04290208
Title: A Comparison of IV Versus PO Acetaminophen Postoperatively for Opioid Consumption After Cesarean Section
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Main Line Health (Other)
Collaborators: Sharpe-Strumia Research Foundation (Other)
Responsible Party: Principal Investigator, Dmitri Chamchad, Anesthesia Research Director, Main Line Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: F/N-R19-3892BLP
Record Dates: First submitted 2019-08-14; First posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Postoperative Pain; Cesarean Section; Acetaminophen
Keywords: Humans; Female; Pregnancy; Acetaminophen; Narcotics; Patient Satisfaction; Cesarean Section; Pain; Postoperative Period
MeSH Terms: conditions — Pain, Postoperative; Patient Satisfaction; Pain | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: When the Principal Investigator calls to enroll patient into the study, pharmacy will be responsible for labelling and delivering the drugs to the labor and delivery unit. The label will include the patient enrollment number and the study name. The investigators will be blind to the patient's drug/placebo assignment. In case of emergency, side effects, or allergic reaction, the pharmacy will be contacted to unblind medication.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous Administration of Acetaminophen (Active Comparator): A single peri-operative dose of acetaminophen 1000 mg IV over 15 minutes after skin is closed.
  Interventions: Drug: Acetaminophen; Drug: Placebos
- Per Oral Administration of Acetaminophen (Active Comparator): A pre-operative liquid dose of acetaminophen 1000mg orally in the on-call to Operative Room.
  Interventions: Drug: Acetaminophen; Drug: Placebos

INTERVENTIONS:
Drug: Acetaminophen — IV Acetaminophen
  Other Names: Tylenol
  Arms: Intravenous Administration of Acetaminophen
Drug: Acetaminophen — Acetaminophen liquid syrup
  Other Names: Tylenol
  Arms: Per Oral Administration of Acetaminophen
Drug: Placebos — Flavored, non-medicated (placebo) liquid syrup
  Other Names: Placebo for acetaminophen
  Arms: Intravenous Administration of Acetaminophen
Drug: Placebos — IV salt solution (non-medicated)
  Other Names: Placebo for acetaminophen
  Arms: Per Oral Administration of Acetaminophen

SUMMARY:
This randomized controlled study will compare narcotic consumption between two groups: patients that receive a perioperative dose of IV acetaminophen versus patients that receive a perioperative dose of oral liquid acetaminophen for scheduled cesarean section.

DETAILED DESCRIPTION:
"Enhanced recovery" is an alternate management protocol described by a multi-modal, evidence based approach to peri-operative care, with the goal of accelerating recovery and return to normal activity after surgery. Results have shown stable pain control with a decrease in narcotic consumption, a quicker return of bowel function, and decreased length of hospital stay and cost with no change in level of patient satisfaction, morbidity, or readmission rate. An aspect of some alternate management protocols is the administration of acetaminophen.

The concentration of acetaminophen in cerebrospinal fluid (CSF) is directly proportional to the analgesic activity of acetaminophen. Acetaminophen relies on a high concentration gradient from the plasma to the CSF in order to passively diffuse into the central nervous system (CNS), its principal site of action. A 2012 study, comparing plasma and CSF pharmacokinetics of intravenous (IV), oral (PO), or rectal (PR) acetaminophen, concluded that IV administration of acetaminophen results in higher plasma and CSF concentration values. Therefore, IV acetaminophen produces better CNS penetration compared to PO or PR methods.

ELIGIBILITY:
Inclusion Criteria:

* Women age 18 or older
* Scheduled to undergo a cesarean section

Exclusion Criteria:

* Existing diagnosis of chronic pain
* Need to undergo a vertical skin incision
* Aspartate Aminotransferase (AST) > 50, alanine aminotransferase (ALT) > 70
* Platelets below 80,000 on admission
* Need to undergo general anesthesia
* Tubal ligation at time of Cesarean section
* Prior or known allergy to any of the medications being utilized in this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2019-08-22 (Actual); Primary Completion 2020-06-23 (Estimated); Study Completion 2020-06-23 (Estimated)

PRIMARY OUTCOMES:
Narcotic Utilization | 6 hours post operative
  The Center for Disease Control and Prevention Morphine Milligram Equivalent Score will be used to calculate total narcotic use (conversion factor for administered opioid x milligrams administered) while the patient remains as an inpatient.

SECONDARY OUTCOMES:
Post-operative Pain Level | Every hour for six hours post-op
  Pain will be measured via the visual analog Postoperative Pain Scale and gathered by nursing. The visual analogue Postoperative Pain Scale indicates the level of pain the patient is feeling or felt in the indicated period from 0 (no pain) to 100 (the worst pain possible).
Patient Satisfaction | Up to 24 hours
  Patient satisfaction will be assessed using the validated survey used in the Mayo Clinical Trial.
Postoperative complications during the inpatient stay | Up to 24 hours
  Postoperative complications will be noted during the inpatient stay.

CONTACTS AND LOCATIONS:
Overall Officials: Dmitri Chamchad, MD, Principal Investigator — Main Line Health; Robert Day, MD, Principal Investigator — Bryn Mawr Hospital
Locations (1):
- Lankenau Medical Center, Wynnewood, Pennsylvania, United States

REFERENCES:
- [Background] Nelson G, Kalogera E, Dowdy SC. Enhanced recovery pathways in gynecologic oncology. Gynecol Oncol. 2014 Dec;135(3):586-94. doi: 10.1016/j.ygyno.2014.10.006. Epub 2014 Oct 12. PMID 25316179
- [Result] Singla NK, Parulan C, Samson R, Hutchinson J, Bushnell R, Beja EG, Ang R, Royal MA. Plasma and cerebrospinal fluid pharmacokinetic parameters after single-dose administration of intravenous, oral, or rectal acetaminophen. Pain Pract. 2012 Sep;12(7):523-32. doi: 10.1111/j.1533-2500.2012.00556.x. Epub 2012 Apr 24. PMID 22524979